CLINICAL TRIAL: NCT00353379
Title: Pharmacology of Cognition in Schizotypal Personality Disorder: Guanfacine for Cognitive Symptoms in Schizotypal Personality Disorder
Brief Title: Pharmacology of Cognition in Schizotypal Personality Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 95-0650; R01MH056140 (NIH); DATR A3-NSS
Record Dates: First submitted 2006-07-14; First posted 2006-07-18 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Schizotypal Personality Disorder; Personality Disorders
MeSH Terms: conditions — Schizotypal Personality Disorder; Personality Disorders | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- guanfacine (Experimental): Participants will take guanfacine.
  Interventions: Drug: Guanfacine
- placebo (Placebo Comparator): Participants will take placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine — Participants will take guanfacine for 6 weeks. Guanfacine dosages will not exceed 2 mg per day.
  Arms: guanfacine
Drug: Placebo — Participants will take placebo for 6 weeks.
  Arms: placebo

SUMMARY:
This study will determine the effectiveness of guanfacine in improving cognitive and functional impairments in schizotypal personality disorder.

DETAILED DESCRIPTION:
Schizotypal personality disorder is a psychiatric condition that is characterized by deficiencies in interpersonal relationships and disturbances in thought patterns, appearance, and behavior. This disorder is different from schizophrenia. While some of the symptoms of the two disorders are similar, such as the tendency to have unusual beliefs and behaviors, people with schizotypal personality disorder do not experience hallucinations and are not significantly disconnected from reality, both of which are signature symptoms of schizophrenia. Guanfacine is a drug that is often used to treat high blood pressure and attention deficit hyperactivity disorder. There is evidence that guanfacine enhances cognition and diminishes impulsivity. This study will determine the effectiveness of guanfacine in improving symptoms of schizotypal personality disorder.

Participants in this 6-week, double-blind study will be randomly assigned to receive either guanfacine or placebo. Participants receiving guanfacine will remain on the drug for the duration of the study. The other participants will receive placebo for the duration of the study. Guanfacine dosages will not exceed 2 mg per day. All participants will report to the study site weekly for assessments of vital signs, study compliance, medication side effects, and psychological symptoms. Additional cognitive testing will be performed at week 6. Upon study completion, patients will return for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male or female
* Medically and neurologically healthy (Medically healthy means that the patient does not have a major or partially treated medical condition that based on the judgment of the research clinician would either put the patient at increased risk and/or affect our findings. Common conditions include: high blood pressure, diabetes, uncontrolled asthma or COPD, abnormal heart rhythm, chronic viral infections. Neurologically healthy means that the patient has not experienced brain injury or head trauma associated with prolonged (e.g., > 10 minutes) loss of consciousness, seizures or other conditions based on the research clinician's judgment would either put the patient at increased risk and/or affect our findings.)
* Between 18 and 60 years of age
* Patients must also be medication free (at least 2 weeks) while participating in guanfacine, except for the following medications: NSAIDS (eg, Advil), Tylenol, Levothyroxine (if on stable dose for 1 month, no symptoms of hypothyroidism and normal thyroid labs), Non-centrally acting antihistamines, H2 blockers (eg, Zantac), PPIs (eg, Prilosec, Prevacid). Research physician will make judgment on case-by-case basis based on risk to subject, and potential confounding effect on data validity.
* Subjects in the SPD group must meet DSM-IV criteria for Schizotypal Personality Disorder.
* Subjects in the AvPD group must meet DSM-IV criteria for Avoidant Personality Disorder and not meet criteria for schizotypal, paranoid, and schizoid personality disorder. In addition, the AvPD group must have fewer than 2 schizotypal traits.

Exclusion Criteria:

* Subjects may not have a significant medical illness (ie, insulin dependent diabetes, gastric/duodenal ulcer), or significant neurological illness (ie epilepsy, CMS, CVA, focal neurological lesion).
* Any cardiovascular condition that, based on the research clinician's judgment (which includes cardiological consultation), would put the participant at increased risk will be considered an exclusion criteria. This would certainly include evidence by history or exam of heart block, tachyarrhythmia, angina, ventricular hypertrophy, those taking antihypertensives. Blood pressure parameters will be a >25% decrease in mean arterial systolic blood pressure from baseline, an orthostatic decrease in systolic blood pressure of 20 mm Hg and/or in diastolic blood pressure of 10 mm Hg, and heart rate parameter will be below 55 bpm.
* Participants are also excluded if they are more than 40% above ideal body weight. The weight limit helps insure that standard doses of guanfacine will not be given to patients who are extremely overweight who might then receive a lower concentration of these drugs in their central nervous system.
* Subjects must also have a corrected or uncorrected visual acuity of 20/40 or better.
* All participants meeting DSM IV criteria for any current or past history of sustained IV-substance dependence are excluded from the study.
* Participants must be free of substance abuse for at least six months.

Healthy Controls:

Inclusion Criteria:

* Healthy control subjects will be selected according to criteria noted in methods, and in age distribution comparable to our patients.
* Healthy controls will be matched to patients on gender and parental socioeconomic status.
* Healthy controls must be male or female between the ages of 18 and 60.

Exclusion criteria:

* for medical illness are identical to those of patients
* must not meet criteria for a current or lifetime DSM-IV diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, or any Axis II disorder.
* a current Axis I or II diagnosis or a family history of psychotic disorder will also be excluded. However, to avoid a group of HC's too highly groomed and unrepresentative of the general population we will not exclude HC subjects meeting criteria for a past Axis I diagnosis, such as adjustment disorder, dysthymic disorder, depressive disorder not otherwise specified, specific phobia, and sleep disorders. In addition subjects meeting criteria for a non-IV substance abuse disorder more than 6 months prior to enrollment will not be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 1995-09 (Actual); Primary Completion 1997-05 (Actual); Study Completion 1997-05 (Actual)

PRIMARY OUTCOMES:
Performance on tests of sustained attention, episodic memory, and working memory | Measured at Week 1
Performance on tests of sustained attention, episodic memory, and working memory | Measured at Week 4

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | Measured at Week 1
Hamilton Depression Rating Scale | Measured at Week 2
Hamilton Depression Rating Scale | Measured at Week 3
Hamilton Depression Rating Scale | Measured at Week 4
Hamilton Depression Rating Scale | Measured at Week 5
Positive and Negative Symptom Scale | Measured at Week 1
Positive and Negative Symptom Scale | Measured at Week 2
Positive and Negative Symptom Scale | Measured at Week 3
Positive and Negative Symptom Scale | Measured at Week 4
Positive and Negative Symptom Scale | Measured at Week 5
Clinical Global Impression Scale | Measured at Week 1
Clinical Global Impression Scale | Measured at Week 2
Clinical Global Impression Scale | Measured at Week 3
Clinical Global Impression Scale | Measured at Week 4
Clinical Global Impression Scale | Measured at Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Larry J. Siever, MD, Principal Investigator — Bronx VA Medical Center/Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] McClure MM, Barch DM, Romero MJ, Minzenberg MJ, Triebwasser J, Harvey PD, Siever LJ. The effects of guanfacine on context processing abnormalities in schizotypal personality disorder. Biol Psychiatry. 2007 May 15;61(10):1157-60. doi: 10.1016/j.biopsych.2006.06.034. Epub 2006 Sep 1. PMID 16950221